CLINICAL TRIAL: NCT07222475
Title: Writing Relaxing Beats in Adolescents Who Have Sickle Cell Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, C. Robert Bennett, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-007609
Record Dates: First submitted 2025-10-27; First posted 2025-10-30 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-10

CONDITIONS: Sickle Cell Disease
Keywords: Music Therapy
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Music Therapy (Experimental): Songwriting intervention
  Interventions: Behavioral: Songwriting intervention (active music therapy)

INTERVENTIONS:
Behavioral: Songwriting intervention (active music therapy) — Participants will engage in a songwriting intervention with a music therapist.

SUMMARY:
This research aims to see if songwriting can help reduce anxiety in adolescents with Sickle Cell Disease. The purpose of the study is to discover if participants find songwriting and playing their songs to be practical and acceptable, and helpful for managing anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 11-18 years of age at the time of enrollment and able to provide assent
* Diagnosed with any type of sickle cell disease
* Currently receiving care at pediatric center
* Able to read and write in English

Exclusion Criteria:

* Care transitioned to adult facility
* Visual, hearing, or cognitive impairment which may impede the ability to complete the songwriting intervention or data collection measures

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in State-Trait Anxiety Inventory score | Baseline, 3 months
  The State and Trait Anxiety Inventory measures anxiety. Participants respond to 20 questions about how they are currently feeling on a 4-point Likert scale of 1 (not at all) to 4 (very much so). A total score is calculated by summing the item responses and ranges from 20 to 80. Higher scores indicate higher anxiety (a worse outcome) and lower scores indicate less anxiety (a better outcome).
Change in Patient Health Questionnaire (PHQ-A) score Change in Patient Health Questionnaire for Adolescents (PHQ-A) score | Baseline, 3 months
  The Patient Health Questionnaire for Adolescents (PHQ-A) is a modified version of the PHQ-9 to be used with adolescents. Participants respond to 9 questions scored on a 4-point Likert scale of 0 (Not at all) to 3 (Nearly every day). A total score is calculated by summing the item responses and ranges from 0 to 27; higher scores are associated with higher levels of or more severe depression.
Change in Connor Davidson Resilience Scale (CD-RISC 10) score | Baseline, 3 months
  The Connor-Davidson Resilience scale (CD-RISC) measures resilience. Participants respond to 10 questions scored on a 5-point Likert scale of 0 (Not true at all) to 4 (True nearly all the time). A total score is calculated by summing the item responses and ranges from 0 to 40; with higher scores reflecting greater resilience.
Change in Difficulties in Emotion Regulation Scale (DERS-SF) score | Baseline, 3 months
  The Difficulties in Emotion Regulation Scale Short Form (DERS-SF) measures difficulties in emotion regulation in adults and adolescents. It consists of six subscales: Nonacceptance, Goals, Impulse, Awareness, Strategies, and Clarity, each with three items. Participants respond to 18 questions scored on a 5-point Likert scale of 1 (Almost never) to 5 (Almost always). A total score is calculating by summing the item responses and ranges from 18 to 90; higher scores indicate greater difficulty with emotion regulation skills.
Change in PROMIS Pediatric Pain Behavior (SF-8a) score | Baseline, 3 months
  The PROMIS Pediatric Pain Behavior (SF-8a) short form measures behaviors that typically indicate to others that an individual is experiencing pain. Participants respond to 8 questions scored on a 6-point Likert scale of 1 (Had no pain) to 6 (Almost always). A total score is calculated by summing the item responses and ranges from 8 to 48, with higher scores indicating a more pain related behavior.
Change in PROMIS Pediatric Pain Quality - Affective (SF-8a) score | Baseline, 3 months
  The PROMIS Pediatric Pain Quality- Affective (SF-8a) short form assesses the emotional distress that accompanies pain. Participants respond to 8 yes or no questions (0 = no, 1 = yes). A total score is calculated by summing the item responses and ranges from 0 to 8, with higher scores indicating a greater impact of pain on emotional distress.
Change in PROMIS Pediatric Pain Quality - Sensory (SF-8a) score | Baseline, 3 months
  The PROMIS Pediatric Pain Quality - Sensory (SF-8a) short form assesses the sensory experiences of pain. Participants respond to 8 questions scored on a 5-point Likert scale of 1 (Not at all) to 5 (Very much). A total score is calculated by summing the item responses and ranges from 8 to 40, with higher scores indicating participants experiencing increased sensory responses to pain.
Change in PROMIS Pediatric Physical Stress Experiences (SF-8a) score | Baseline, 3 months
  The PROMIS Pediatric Physical Stress Experiences (SF-8a) short form assess the physically experienced sensations associated with pain. Participants respond to 8 questions scored on a 5-point Likert scale of 1 (Never) to 5 (Always). A total score is calculated by summing the item responses and ranges from 8 to 40, with higher scores indicating a greater impact of pain on physical stress experienced.
Change in PROMIS Pediatric Psychological Stress Experience (SF) score | Baseline, 3 months
  The PROMIS Pediatric Psychological Stress Experience (SF) short form assesses the thoughts and feelings associated with pain. It measures facets of stress, including feeling overwhelmed, lack of perceived control, and cognitive-perceptual disruption, using a 7-day recall period. Participants respond to 8 questions scored on a 5-point Likert scale of 1 (Never) to 5 (Always). A total score is calculated by summing the item responses and ranges from 8 to 40, with higher scores indicating a greater impact of pain on psychological stress.
Change in PROMIS Pediatric Physical Activity (SF) score | Baseline, 3 months
  The PROMIS Pediatric Physical Activity (SF) measure self-reported capability of physical activities. Participants respond to 8 questions scored on a 5-point Likert scale of 0 (No days) to 5 (6-7 days). A total score is calculated by summing item responses and ranges from 0 to 40, with higher scores indicating a greater deal of physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: C. Robert Bennett, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Division of Nursing, Rochester, Minnesota, United States